CLINICAL TRIAL: NCT04474977
Title: Microvascular Decompressive Surgery for Hemifacial Spasm: Nuances of Technique and Outcome
Brief Title: Microvascular Decompressive Surgery for Hemifacial Spasm
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Zanaty, Asisstant Lecturer, Assiut University
Other Study IDs: Hemifacial Spasm
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Hemifacial Spasm
MeSH Terms: conditions — Hemifacial Spasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Microvascular Decompressive Surgery — Microvascular decompression for hemifacial spasm

SUMMARY:
* Review the clinical outcomes of Micro vascular decompression of Hemi facial Spasm.
* Assess safety and efficacy of Micro vascular decompression.
* Improve the outcome of these patients and decease rate of recurrence and complications.

DETAILED DESCRIPTION:
Hemi facial spasm (HFS), a term described in 1905 by Babinski but first reported by Schultz in 1875, is a highly morbid movement disorder characterized by intermittent involuntary movement of muscles innervated by the facial nerve.

(HFS) affects roughly 10 in 100,000 individuals in fifth or sixth decades of life.

Primary HFS is commonly attributed to vascular loops compressing the seventh cranial nerve at its exit zone from the brainstem. The facial nerve compression is thought to lead to ephaptic transmission and to hyperactivity of the facial nucleus, resulting in the involuntary facial movements.

Secondary HFS frequently follows peripheral facial palsy or may arise from facial nerve damage produced by tumours, demyelinating disorders, traumatisms, and infections accounting for 1-2 & of HFS.

Over four in five primary HFS cases involve either anterior or posterior inferior cerebellar artery as the primary offender although vertebral artery, multiple vessels and veins may be involved.

EMG recordings confirm the diagnosis by showing a typical electrophysiological signature: clonic facial muscle contractions, hyperactivity, and synkinesis, lateral spread evoked responses.

Imaging can be useful for confirming that HFS is primary in nature and due to a neurovascular compression. In most cases (95% of the patients) the compressive vessel, generally an artery, is seen on MRI combined with MR-Angiography (MRA). High resolution T2-sequence is to be used to get good delineation of the facial nerve.

Many treatments for HFS have been reported, including pharmacological agents, botulinum toxin injection, facial nerve blockage, physical therapy, radiofrequency ablation, acupuncture, as well as facial nerve combing and microvascular decompression (MVD).

However, while MVD is effective, there are still significant postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

Primary Hemi facial spasm Unilateral Adults 20-60 years Clinical Diagnosis confirmed by Facial Evoked potential & Neuroimaging

Exclusion Criteria:

Secondary Hemi facial spasm caused by intracranial masses or other lesions Recurrent Hemi facial spasm Patients who are unfit for any neurosurgical interventions.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The sample size calculated by sample size calculator software according to:
  1. confidence interval : 95%
  2. power : 80%
  3. P-value : 5%
  4. Prevalence : 0.79/100000
  5. Population size: 110,000 referenced by Assiut health directory statistics 2018 All cases that fulfil the selection criteria that will be admitted in the department of neurosurgery at Assiut university hospital with expected size of at least 30 patients
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Samsung Medical center Grading system for Severity of Hemifacial Spasm | one month
  Success rate by assessing the degree of hemifacial spasm pre and post-operative using the SMC grading system proposed by Lee et all
Hearing Affection | one month
  Audiometry: to detect the degree of post-operative hearing affection using WHO Grading system For Hearing Loss
Recurrence | Six Month
  Recurrence rate within the duration of follow up
Morbidity and mortality | Six Month
  Morbidity and mortality rates related to the procedure using modified Rankin Scale

SECONDARY OUTCOMES:
changes in facial evoked EMG | one month
  Detect the changes in facial evoked EMG preoperative and postoperative and its correlation to outcomes (esp. disappearance of lateral spread response)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] THUREL R. [Peripheral facial hemispasm, trigeminal neuralgia and masticatory spasm on the same side]. Rev Neurol (Paris). 1951;85(4):288-9. No abstract available. Undetermined Language. PMID 14921388
- [Background] Wu Y, Davidson AL, Pan T, Jankovic J. Asian over-representation among patients with hemifacial spasm compared to patients with cranial-cervical dystonia. J Neurol Sci. 2010 Nov 15;298(1-2):61-3. doi: 10.1016/j.jns.2010.08.017. PMID 20864122
- [Background] Auger RG. Hemifacial spasm: clinical and electrophysiologic observations. Neurology. 1979 Sep;29(9 Pt 1):1261-72. doi: 10.1212/wnl.29.9_part_1.1261. PMID 573406
- [Background] Cui Z, Ling Z. Advances in microvascular decompression for hemifacial spasm. J Otol. 2015 Mar;10(1):1-6. doi: 10.1016/j.joto.2015.06.002. Epub 2015 Jul 26. PMID 29937774
- [Background] Hyun SJ, Kong DS, Park K. Microvascular decompression for treating hemifacial spasm: lessons learned from a prospective study of 1,174 operations. Neurosurg Rev. 2010 Jul;33(3):325-34; discussion 334. doi: 10.1007/s10143-010-0254-9. Epub 2010 Mar 27. PMID 20349099
- [Result] Sindou M, Mercier P. Microvascular decompression for hemifacial spasm: Outcome on spasm and complications. A review. Neurochirurgie. 2018 May;64(2):106-116. doi: 10.1016/j.neuchi.2018.01.001. Epub 2018 Feb 15. PMID 29454467